Fundação Bahiana de Infectologia
CNPJ: 02.340.960/0001-26
Rua João das Botas, 185, Salas 703-705,
Canela, 40110-160, Salvador-Bahia.
Telefone: +55 (71) 3247-2756

TITLE: IMPACT OF A DOLUTEGRAVIR-BASED REGIMEN ON EARLY MORTALITY OF SEVERELY IMMUNOCOMPROMISED AIDS PATIENTS: A PILOT STUDY

NCT number: NCT01837277

Date: 20 June 2018

# **Statistical Analysis Plan**

#### **General Considerations**

All abstracts and statistical analyzes will be provided for the intended **intention to treat population**, defined as all participants who are randomized to treatment. With the exception of the Primary Efficacy Parameter Analysis, percentage of responders for the intent-to-treat population, missing data will not be estimated or transported in any statistical analyzes.

All comparisons of treatment groups will be performed using two-tailed tests at a significance level of 0.05 (p <0.05). The null hypothesis for all analyzes is that there is no difference between the treatment groups.

All abstracts, statistical analyzes and individual record data of participants described below will be provided in separate annexes. Separate listings will be provided for each of the treatment groups in the intention-to-treat population.

## **Arrangement of participants**

Summaries of the number of randomized patients, number of those completing the study, and incidence of protocol violations will be provided for each treatment group. The number (%) of participants with protocol violations that may affect study objectives will be based on database analysis. This evaluation will be done before determining the allocation of treatment for all participants in the database.

## **Demographic Characteristics and Disease**

The statistical analyzes described below will be completed to:

- The population of intention to treat participant:
- The evaluable population of effectiveness.

Demographic Characteristics

The table below identifies the demographic and disease characteristics used to determine the comparability of treatment groups and the methods used to analyze them.

Table 1 - Variables analyzed to determine comparability

| Variable | Analysis method |
|-------------|-----------------|
| Basal age | One-way |
| | ANOVA/KW |
| Basal VL | One-way |
| | ANOVA/KW |
| CD4 + basal | One-way |
| | ANOVA/KW |

The primary efficacy endpoint is the number (%) of participants who achieved the primary endpoint (HIV-1 Viral Load RNA <50 copies / ml) at week 48 (or discontinuation) visit. Participants will be counted as non-responders if they do not attend Week 48 (or term).

The DTG treatment group will be compared to the EFV group with respect to the percentage of responders using a chi-square test. Two-tailed, 95% confidence intervals for the percentage of responders will be calculated for each treatment group.

The following table identifies the secondary endpoints of effectiveness and the methods used to analyze them.

Table 2 - Variables analyzed in the main points of analysis

| Variable | Analysis method |
|---------------------------------------------|-----------------|
| Frequency of Adverse Events | chi-square test |
| Proportion of participants achieving VL <50 | chi-square test |
| copies / ml at each point of analysis | |
| Proportion of deaths | chi-square test |

| CD4 + count at each point of analysis | One-way ANOVA/KW |
|---------------------------------------|------------------|
|---------------------------------------|------------------|

## **Security Endpoints**

Summaries and statistical analyzes of safety parameters will be completed for the population by intention to treat. The incidence of at least one grade III or IV event will be the primary safety objective of the study. Treatment groups will be compared to the percentage of participants with at least one grade III or IV adverse event using a Chisquare test.

### **Serious Adverse Events**

Secondary safety endpoints are the incidence of adverse events classified according to the preferred term and body system, the results of clinically significant laboratory tests and changes in vital signs. Treatment groups will be compared with the percentage of participants with clinically significant laboratory test results at Week 4, 8, 16, 24, 36 or 48 visits using Chi-square.

Summaries of physical examination data, vital signs (actual value and baseline change) and laboratory data (real value and change of baseline) will be provided at each visit.

#### **Report of Adverse Experiences**

The investigator and local staff will be responsible for documenting, detecting and reporting events that correspond to the definition of Adverse Event, which is defined as any undesired medical event occurring in a participant or individual involved in a clinical investigation protocol, which may be transiently associated with the use of a medical product, whether or not it is considered to be related to the test product. A serious adverse event (SAE) is defined as any medical event that results in death or life-threatening, hospitalization, disability, congenital anomaly, or all grade 3 or higher liver damage caused by drugs.